CLINICAL TRIAL: NCT03047486
Title: Smartguard Use in Real Life : a Longitudinal Study in Patients With Type 1 Diabetes
Acronym: Smartguard
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 16-106
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2017-02

CONDITIONS: Type 1 Diabetes Mellitus Maturity Onset
Keywords: insulin pump; continuous glucose monitoring sensor; predictive low glucose suspend

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The reference treatment of the type 1 diabetes is intensified insulin therapy by insulin pump. The CGM (continuous glucose monitoring) is a technology available for a decade, which allows the continuous measure of interstitial glucose rate. The results are available in real time to the user, who can so use them to optimize the adjustment of its treatment by insulin pump. Since a few years, several research programs aim for finalizing an automated system using the data of real time interstitial glucose to adjust automatically, via an algorithm, the release of insulin by the pump. This type of closed-loop system is for the moment only experimental, not still widely available in routine. On the other hand, rudimentary regulation systems partially automated already exist and can be used in common clinical practice. One of these systems, Smartguard ®, allows this type of regulation to decrease the hypoglycemic risk of the patients treated by insulin pump. It is indeed a hypo minimizer which interrupts the basal output when the algorithm embarked on the pump determines thanks to the CGM data what a hypoglycemia risks to occur in the 30 minutes. The efficiency of this system to reduce hypoglycemias was proved by several studies in pediatric and adult populations of subjects with DT1 (Diabetes Care on 2015; 38:1197-1204. J Diabetes Sci Technol. 2016 May 20. Pii: 1932296816645119). However, to date, there are no published data concerning the method of use of this system (sensor et pump initial configuration; patient education), nor the evolution of the sensor and pump parameters during the use.

The aim of this observationnelle study is to collect the data of efficiency, safety and use of the system Smartguard ® in common clinical practice in an adult population of subjects DT1.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes ≥ 1 year
* CSII ≥ 6 months
* Previous education to flexible insulin therapy
* Patient willing to use sensors and smartguard option for 1 year
* A1c ≥ 7.5% and/or severe hypoglycemia ≥ 2 episodes during the last 6 month and/or recurrent hypoglycemia and/or hypoglycemia unawareness and/or brittle diabetes

Exclusion Criteria:

* No access to a computer and/or to the web making it impossible to follow patients through telemedicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective trial involved adult patients with Type 1 Diabetes for at least 1 year, and a treatement by insulin pump (CSII) for at least 6 months, to study and describe the efficacy and safety of the predictive low glucose suspend (PLGS) system in real life, in difficult diabetes (severe hypoglycemia, unawared hypoglycemia, brittle diabetes).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Glucose TIR (time in range) from CGM recording | change between baseline and after 12 month
  TIR will be calculated from the CGM recording, thanks to the medtronic carelink software
Glucose Time below range (hypoglycemia < 70 mg/dl) from CGM recording | change between baseline and after 12 month
  Time below range will be calculated from the CGM recording, thanks to the medtronic carelink software

SECONDARY OUTCOMES:
HbA1c | month 0, 3, 6, 9, 12

OTHER OUTCOMES:
daily insulin total dose | month 0, 3, 6, 9, 12
basal / bolus ratio | month 0, 3, 6, 9, 12
daily bolus number | month 0, 3, 6, 9, 12
Mean daily hypoglycemic predictive-stop time | month 0, 3, 6, 9, 12
Mean daily hypoglycemic-stop time | month 0, 3, 6, 9, 12
Time Percentage with CGM Sensor Use Time | month 0, 3, 6, 9, 12
Medical time at each consultation | month 0, 3, 6, 9, 12

CONTACTS AND LOCATIONS:
Overall Officials: Michael JOUBERT, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- Endocrinology Unit and Clinical Research Center Basse Normandie, University Hospital of Caen, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joubert M, Briant AR, Kessler L, Fall-Mostaine F, Dubois S, Guerci B, Schoumacker-Ley L, Reznik Y, Parienti JJ. Sensor-Augmented Insulin Pump with Predictive Low-Glucose Suspend (PLGS): Determining Optimal Settings of Pump and Sensor in a Multicenter Cohort of Patients with Type 1 Diabetes. Diabetes Ther. 2022 Sep;13(9):1645-1657. doi: 10.1007/s13300-022-01302-3. Epub 2022 Aug 1. PMID 35913656